CLINICAL TRIAL: NCT01958632
Title: Evaluation of Sensory Recovery After Reconstruction of Digital Nerves of the Hand Using Muscle-in-vein Conduits in Comparison to Nerve Suture or Nerve Transplantation
Brief Title: Muscle-in-vein Conduits for Digital Nerve Reconstruction
Status: Completed | Type: Observational
Sponsor: BG Trauma Center Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Theodora Manoli, M.D., Plastic Surgeon, BG Trauma Center Tuebingen
Other Study IDs: 117/2012BO2
Record Dates: First submitted 2013-10-05; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Sensory Recovery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- N: nerve suture
  Interventions: Procedure: Nerve reconstruction
- NT: nerve transplantation
  Interventions: Procedure: Nerve reconstruction
- VM: vein-in-muscle conduit
  Interventions: Procedure: Nerve reconstruction

INTERVENTIONS:
Procedure: Nerve reconstruction

SUMMARY:
The actual study should provide a first direct comparison between results after reconstruction of sensory nerves of the hand using muscle-in-vein conduits to the standard methods of nerve transplantation and direct nerve suture.

ELIGIBILITY:
Inclusion Criteria:

complete digital nerve injuries, nerve reconstruction in the first 6 months post trauma

Exclusion Criteria:

total or subtotal amputations

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Semmes-Weinstein-Monofilament test | The earliest 6 months post-OP

SECONDARY OUTCOMES:
Two-point-discrimination | The earliest 6 months post-OP

CONTACTS AND LOCATIONS:
Locations (1):
- BG Trauma Center, Tübingen, Germany